CLINICAL TRIAL: NCT07263074
Title: Feasibility and Preliminary Efficacy of a Digital Story Intervention to Facilitate Decision-Making in Patients With Myeloid Cancers Considering Allogeneic Hematopoietic Cell Transplantation
Brief Title: Considering alloHCT: Opportunities for Patient Reflection During Decision-Making Via Digital Stories
Acronym: CHORDS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Rachel Rodenbach, Assistant Professor - Department of Medicine, Hematology/Oncology (SMD), University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UOCPC25049
Record Dates: First submitted 2025-11-17; First posted 2025-12-04 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Myeloid Malignancy

STUDY DESIGN:
Intervention Model Description: Assess the feasibility of CHORDS among patients with myeloid cancers referred for alloHCT.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (CHORDS) (Experimental): The CHORDS intervention consists of 1) digital stories created by individuals who previously underwent consultation for alloHCT and 2) explicit values clarification exercises designed to help patients reflect on their emotions and clarify what matters to them, including a) an interactive workbook, and b) best-worst scaling (BWS).
  Interventions: Other: CHORDS
- Usual Care (No Intervention): Patients randomized to the usual care arm will receive standard of care. Patients (and their caregivers when available) randomized to usual care will not participate in CHORDS. Patients and caregivers will complete baseline (T1) and post-alloHCT office visit (T3, T4, T5) assessments.

INTERVENTIONS:
Other: CHORDS — The CHORDS intervention consists of 1) digital stories created by individuals who previously underwent consultation for alloHCT and 2) explicit values clarification exercises designed to help patients reflect on their emotions and clarify what matters to them, including a) an interactive workbook, and b) best-worst scaling (BWS).
  Arms: Intervention (CHORDS)

SUMMARY:
This is a two-arm pilot randomized trial that assesses the feasibility and preliminary efficacy of a digital story and values clarification intervention (Considering alloHCT: Opportunities for Patient Reflection During Decision-Making via Digital Stories [CHORDS]) compared to usual care among patients with myeloid cancers considering allogeneic hematopoietic cell transplantation (alloHCT).

DETAILED DESCRIPTION:
Our proposed intervention is Considering alloHCT: Opportunities for Patient Reflection During Decision-Making via Digital Stories (CHORDS), which includes: 1) real-life digital stories of individuals with similar experiences who previously underwent consultation for allogeneic hematopoietic cell transplantation and their caregivers and 2) explicit values clarification exercises designed to help patients reflect on their emotions and clarify what matters to them, including a) an interactive workbook, and b) best-worst scaling. Together, they help patients reflect on their values and prioritize their own needs and goals, enhance emotional awareness, and gain experiential knowledge from peers to better understand the real-life implications of treatment risks and benefits.

ELIGIBILITY:
Patients

Inclusion criteria:

1. Age >21 years old
2. Diagnosis of myeloid cancer (AML, MDS, myelofibrosis, CML, or MDS/MPN)
3. Being considered for alloHCT
4. Able to provide informed consent
5. Able to speak English. The reason for this is because the digital stories have been created in the English language and their multimedia form cannot easily be translated.

Exclusion criteria 1) Patients with psychiatric or cognitive conditions which the hematologist believes prohibits informed consent or compliance with study procedures

Caregivers

Inclusion criteria:

1. Age >18 years old
2. Selected by the patient when asked if there is a "family member, partner, friend or caregiver with whom you discuss or who can be helpful in health-related matters."
3. Caregiver may be paid/professional or informal caregiver
4. Able to provide informed consent
5. Able to speak English

Exclusion Criteria:

1) None

Hematologists

Inclusion criteria:

1) Hematologists of the patients who agree to enroll on the study who are part of Wilmot Cancer Institute.

Exclusion criteria

1) None

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-01-15 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Retained (Feasibility - Retention Rate) | From enrollment (Day -30 to Day 0) to 2 weeks post-alloHCT office visit (Day 9-19)
  Feasibility will be assessed based on the percentage of enrolled participants who complete both the intervention and post-intervention secondary outcome assessments. The number of participants who complete all study procedures will be divided by the total number enrolled to calculate the retention rate. Higher percentages indicate greater feasibility.

SECONDARY OUTCOMES:
Mean Change in Decisional Engagement Scale Score | Baseline (Day -30 to Day 0) to 2 weeks post-alloHCT office visit (Day 9-19)
  Engagement in decision making will be assessed using the Decisional Engagement Scale, a self-reported measure evaluating patient involvement and perceived shared decision making. A single score will be derived according to scale instructions. Higher scores indicate greater engagement in decision making. There are 10 items in the scale, with each items score ranging from 0 to 10 (range 0-100 for the entire scale).
Mean Change in Decisional Conflict Scale Score | Baseline (Day -30 to Day 0) to 2 weeks post-alloHCT office visit (Day 9-19)
  Decisional conflict will be assessed using the Decisional Conflict Scale, a validated self-report instrument that measures personal uncertainty in making health-related decisions. The total score is derived by averaging item responses according to the scoring manual (range 0-100). Higher scores indicate greater decisional conflict (worse outcome), while lower scores indicate less conflict (improvement).
Mean Change in Distress Thermometer Score | Baseline (Day -30 to Day 0) to 2 weeks post-alloHCT office visit (Day 9-19)
  Psychological distress will be measured using the NCCN Distress Thermometer, a single-item visual analog scale ranging from 0 ("no distress") to 10 ("extreme distress"). Higher scores indicate greater distress.

OTHER OUTCOMES:
Qualitative Analysis of Patient-Hematologist Discussion of Values and Goals | Following alloHCT office visit (Day 9 to 194)
  Audio recordings of alloHCT office visits will be transcribed and analyzed using qualitative methods to identify the presence and nature of discussions related to patient values and treatment goals.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No